CLINICAL TRIAL: NCT06412796
Title: Comparison of Postoperative Analgesic Effectiveness of Subcostal Transversus Abdominis Plane Block Versus External Oblique Intercostal Block on Patients With Gastric Cancer Undergoing Gastrectomy
Brief Title: Postoperative Analgesic Effects of Subcostal Transversus Abdominis Plane Block Versus External Oblique Intercostal Block on Patients Undergoing Gastrectomy
Status: Not yet recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayse Ulgey, Professor Doctor, TC Erciyes University
Other Study IDs: 2023/600
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain; Analgesia
Keywords: SCTAP; External Oblique Intercostal block; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subcostal Transversus Abdominis Plane (SCTAP) block.: SCTAP Block is performing by USG probe positioned on the anterior abdominal wall immediately inferior to the costal margin and then needle advanced to 2 to 3 cm lateral to the aponeurosis of the external oblique muscles, internal oblique muscles, and transversus abdominis in the TAP. Saline 0.5mL was injected to determine the position of the transverse fascia and 15-20 ml local anesthetics injected both in right and left sides of abdomen.
- External Oblique Intercostal (EOI) block: EOI block is performed by placing the US probe in paramedian sagittal orientation at the T6-7 level and visualizing the external oblique and intercostal muscles. Local anesthetics inject the under the external oblique muscle.

SUMMARY:
Open Gastrectomy surgery is a big surgery with upper umbilical median incision where the postoperative pain is occur frequently. pain managements of this surgery with intravenous opioid analgesics are currently standard approach. but its side effects as sedation, decreased bowel movement and respiratory depression are limiting its use. so local anesthesia done with regional block methods provides good analgesia after surgery that decrease use of opioid analgesics. in this study we intend to compare subcostal TAP block with external oblique intercostal block

DETAILED DESCRIPTION:
in our study, we include the patients who has diagnosed Gastric Cancer and going to open gastrectomy surgery. this surgery performing with initial upper umbilical median incision of abdomen and then removing part or all of the stomach organ, which is cause postoperative pain on all abdominal area and affect the patient's recovery and morbidity. perioperative pain management is also important part of recovery after surgery. intravenous morphine using is part of protocols in analgesics. lately opioid free analgesia is aimed because of opioids side effects such as sedation, respiratory depression and decrease in bowel movement affect patients' recovery and duration in hospital. in this way regional and local anesthetics methods are getting more interested in pain management. To ensure the analgesic effects of the upper umbilical median incision area we planned to perform External Oblique Intercostal (EOI) block and Subcostal Transversus Abdominis Plane (SCTAP) block. To get better results we performed both blocks with Ultrasound Guided Imaging and injected bilateral with 15-20 ml of diluted local anesthetics on each side before the surgery. We divide patients into two groups: Group 1: the patients who get SCTAP block and Group 2: the patients who get EOI block. After the general anesthesia and intubation of patient we clean the abdominal area within antiseptic to perform injection before the surgery is began. In Group 1, SCTAP Block is performing by USG probe positioned on the anterior abdominal wall immediately inferior to the costal margin and then needle advanced to 2 to 3 cm lateral to the aponeurosis of the external oblique muscles, internal oblique muscles, and transversus abdominis in the TAP. Saline 0.5mL was injected to determine the position of the transverse fascia and 15-20 ml local anesthetics injected both in right and left sides of abdomen. In Group 2, EOI block is performed by placing the US probe in paramedian sagittal orientation at the T6-7 level and visualizing the external oblique and intercostal muscles. Local anesthetics inject the under the external oblique muscle. After the surgery patient controlled analgesia (PCA) is given to patients if there will not enough analgesic management confirmed. Pain assessment will be evaluated with the visual pain scale at 2/6/12/24 hours after surgery completed.

ELIGIBILITY:
Inclusion Criteria:

* patients who have diagnosed Gastric Cancer and undergoing Gastric resection
* patients accepted to participate for study

Exclusion Criteria:

* parients that not agreed for the study
* patients who undergoing for second operation at the same surgery incision
* patient that have chronic pains and multiple drugs using
* patients that have psychiatric disorders
* bariatric surgery
* patients with allergics for local anaesthetics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adult patients with gastric cancer who are undergoing gastrectomy and agreed for a study are accepted
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-26 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Need of morphine analgesia | 24 hours
  postoperatively monitoring of patients that need analgesics by morphine consumption using a patient contral analgesics device that record amount of used and wanted analgesics by patients themselves
patients pain scales | 24 hours
  asking patients for pain at postoperative period by visual analog scale and score accordingly

CONTACTS AND LOCATIONS:
Locations (1):
- University of Erciyes, Kayseri, Talas, Turkey (Türkiye)